CLINICAL TRIAL: NCT06781697
Title: InTRavenous kEtAmine and immerSive virtUal Reality to Treat dEpression (TREASURE Trial): a Pilot, Randomized Controlled Trial
Brief Title: InTRavenous kEtAmine and immerSive virtUal Reality to Treat dEpression
Acronym: TREASURE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6159
Record Dates: First submitted 2024-12-19; First posted 2025-01-17 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Treatment Resistant Depression
Keywords: Depression; Ketamine; Virtual Reality; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: A two-phase prospective randomized controlled pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-Ketamine (VR-K) (Experimental): Participants will receive a standard course of ketamine treatment. At the onset of each ketamine therapy session, participants will be provided with an Oculus VR headset, and will be immersed in a tailor-made virtual environment of positive outdoor scenes.
  Interventions: Drug: Ketamine; Device: Oculus VR headset
- Ketamine alone (Active Comparator): Participants will receive a standard course of ketamine treatment.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Standard-of-care ketamine treatment in the outpatient setting: 0.5 mg/kg IV infused over 45 minutes (with monitoring up to 90 minutes) per session, with 2 sessions per week for 2 weeks (total 4 treatments).
Device: Oculus VR headset — Immersion in 45 minutes of virtual environments using the Oculus VR headset during each ketamine infusion.
  Arms: VR-Ketamine (VR-K)

SUMMARY:
Depression is a common condition, with serious negative effects on the health and quality of life of those affected. While there are currently various medications which attempt to treat depression, they often take a long time to begin to work and do not work at all for many people. There is therefore a need for new treatments which work quickly and effectively.

One such medication is called ketamine. Studies have shown that ketamine can treat symptoms of depression quickly. This quick action sets ketamine apart from many antidepressants that take weeks to show noticeable effects. One way that it may do this is by creating a transient sense or feeling of being separated from reality, such as seeing or hearing things that are not really there. Another way to create these same feelings is with virtual reality (VR), where a person can feel as though they are entering a 3-dimensional virtual computer-generated world by wearing a special headset or goggles with a computer inside.

In this study, all participants will receive standard ketamine treatments for depression. Half of the participants will also use a VR headset while receiving the ketamine treatments to see if ketamine and VR acting together provide a better treatment for symptoms of depression than ketamine alone.

This is a small pilot trial. The main purpose of this trial is to learn if it is possible to run a larger clinical trial comparing "ketamine and VR" with "ketamine alone", for adults with treatment-resistant depression. The researchers will study this by seeing how many participants take part in the study within 1-2 years, and how many complete the study treatments and tests. The researchers will also compare the two study groups to see if "ketamine and VR" provide a better treatment for symptoms of depression than "ketamine alone".

DETAILED DESCRIPTION:
Depression is the single largest contributor to global disability, and afflicts individuals of all ages, races, genders, and classes. The significant morbidity is associated with depressive disorders relates to myriad direct and indirect financial costs to individuals and society. It also bears significant mortality, as one of the strongest risk factors for suicide.

Depression is also challenging to treat, with standard antidepressant therapy providing remission to only one third of patients, and incompletely improving the condition of another one third. Even when standard therapy is effective, it can take as long as six weeks for improvement of cognitive/emotional symptoms to become apparent. The final one third of patients often undergo a therapeutic odyssey in which various medications are attempted with no measurable benefit. Ultimately these patients receive a diagnosis of treatment-resistant depression (TRD).

Ketamine has emerged as a fast-acting intervention for the treatment of depressive disorders, which can reach maximum efficacy in only 24 hours and persist for 1-2 weeks. Ketamine is safe, well-tolerated, familiar to many providers and has become widely available as a treatment for depression.

Virtual reality (VR), a technology which immerses users in a controlled digital experience, has also recently been recognized for its potential in the treatment of mental health disorders and recent studies have identified similarities in proposed mechanisms for ketamine and VR in the treatment of depression (e.g. the creation of a non-ordinary and non-rigid experiences of consciousness, and the production of evocative or hallucinatory sensory experiences). However, this combination of interventions has not yet been studied.

Here, the investigators propose to study the combined effect of ketamine and VR in the vulnerable adult mental health population undergoing ketamine therapy for treatment-resistant depression (TRD).

In Phase I of the study, participants (N=3-5) will provide feedback to develop the VR software for this study population.

In Phase II, study participants (N=26) will be randomized to control (standard of care ketamine alone, Group I) or intervention (VR + ketamine concurrently (VR-K), Group II) groups to report on protocol feasibility and to inform the development of a definitive trial to assess VR-K treatment efficacy. All participants will receive a typical sub-anesthetic dose of ketamine (0.5mg/kg) infused intravenously (IV) over 45 minutes, and will be monitored by research staff for up to 90 minutes post-procedure. Each participant will receive a total of 4 ketamine treatments, 2 treatments per week for 2 weeks. All patients will continue their baseline antidepressant regimens while engaged in the study, consistent with standard ketamine therapy for TRD. Participants in the intervention group will wear a virtual reality headset at the onset of each standard ketamine therapy session, and will be immersed in a tailor-made virtual environment of positive outdoor scenes to provide relaxation and reprieve from negative thoughts.

Psychometric surveys will be used to assess the effects of both treatment arms on mood and psychiatric outcomes (depression and anxiety symptoms), side effects (sedation, dissociation, vitals), cognitive function, neural activity (EEG), and patient satisfaction with virtual reality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, able to provide informed consent
* Patient diagnosed with treatment-resistant depression
* Outpatient recommended and approved by psychiatrist for ketamine treatment
* Patients who are on IV ketamine and requiring at least 4 treatments of IV ketamine per course (prescribed by their physiatrist)
* Cognitively alert, oriented, and able to watch immersive content and respond to questions
* Negative human chorionic gonadotropin test before treatment, for female participants of childbearing potential who are not practicing medically appropriate methods of birth control (e.g., hormonal contraceptives, implants, injectables, intrauterine devices, intrauterine systems, etc.)

Exclusion Criteria:

* History of psychosis/comorbid psychiatric disorders/psychotic depression/dissociative syndromes, significant personality disorder, as clinically assessed by psychiatrist
* Using non-prescribed substance (e.g., cannabis) or alcohol use within the preceding 48 hours of treatment
* History of substance misuse and/or dependence, including chronic alcohol abuse
* Previous ketamine use
* Acute dementia/delirium
* Acute risk of suicide at baseline, as determined by the study psychiatrist
* Pregnancy/breastfeeding
* Previous sensitivity to ketamine or related compounds
* Unstable medical condition which may require anesthesia consult
* History of elevated intracranial pressure or cerebrovascular accident
* Recent (within 6 weeks) major cardiovascular event (such as myocardial infarction)
* Significant motion sickness (i.e. occur during exposure to physical/visual and virtual motion, cybersickness, etc.) self-identified by patient
* Inability to communicate with the study team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Number of Participants who Complete at least 90% of Study Follow-ups | From enrolment until the end of follow-ups at 3 months
  The number of participants who achieve at least 90% completion of follow-ups in Phase II will be calculated.
Feasibility - Time Required to Complete Enrolment | At the time of enrolment
  The time required to enrolled to recruit 26 participants in Phase II of the pilot trial will be recorded.

SECONDARY OUTCOMES:
Mood and Psychiatric Outcomes - Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline, 60 minutes and 24 hours after each treatment, and during 1,2,3-week and 1 and 3 month follow-ups
  The MADRS is a 10-item clinician rated scale for measuring severity in the symptoms of depression. Responses for each item are measured on a scale of 0-6 (from no depressive symptomatology to severe depressive symptoms).
Mood and Psychiatric Outcomes - General Anxiety Disorder-7 (GAD-7) | Baseline, 60 minutes and 24 hours after each treatment, and during 1,2,3-week and 1 and 3 month follow-ups
  A self-reported questionnaire measuring severity of symptoms of anxiety. The total score on the GAD-7 ranges from 0 to 21, with 0 indicating no anxiety and 21 indicating severe anxiety.
Mood and Psychiatric Outcomes - Positive and Negative Affect Schedule (PANAS) | Baseline, 60 minutes and 24 hours after each treatment, and during 1,2,3-week and 1 and 3 month follow-ups
  Self-reported assessment of positive and negative emotions. For positive emotions, scores can range from 10-50, with higher scores representing higher levels of positive affect. For negative emotions, scores can range from 10-50, with lower scores representing lower levels of negative affect.
Mood and Psychiatric Outcomes - Patient Health Questionnaire (PHQ-9) | Baseline, 24 hours after each treatment, and during 1,2,3-week and 1 and 3 month follow-ups
  A self-reported 9-item questionnaire to assess degree of depression severity. Total scores can range from 0 to 27, with higher scores indicating more severe depression.
Mood and Psychiatric Outcomes - Beck Depression Inventory-II (BDI-II) | Baseline, 24 hours after each treatment, and during 1,2,3-week and 1 and 3 month follow-ups
  Self-reported questionnaire about symptoms of depression, such as mood, self-dissatisfaction, guilt and fatigue. Scores range from 0 to 63, with higher scores representing higher depression severity.
Anti-depressant use | Baseline, 1 and 3 month follow-ups
  The antidepressant use by participants will be collected.
Ketamine Side Effects - Heart Rate | Before, continuously during the 45-minute infusion, and up to 60 minutes after each treatment
  Heart rate will be collected before, during, and up to 60 minutes after each treatment.
Ketamine Side Effects - Mean Arterial Pressure | Before, continuously during the 45-minute infusion, and up to 60 minutes after each treatment
  Mean arterial blood pressure will be collected before, during, and up to 60 minutes after each treatment.
Ketamine Side Effects - Level of consciousness | At baseline, once during the 45-minute infusion, and up to 60 minutes after each treatment
  Participants' level of consciousness will be assessed using the Observer's Assessment of Alertness/Sedation Scale (OAA/S) to establish whether VR engagement is limited by ketamine's effects. The OAA/S score ranges from 1 to 5, with 1 indicating deep sleep/unconsciousness and 5 indicating alertness.
Ketamine Side Effects - Dissociative Experiences and Psychotomimetic Side Effects | At baseline, 5-10 minutes after the start of each infusion and 60 minutes after each treatment
  The Clinician Administered Dissociative Symptoms Scale (CADSS-6) will be used to assess dissociative experiences and psychotomimetic side effects (i.e., hallucinations, mild depersonalization, derealization, altered time, body perception). Total scores range from 0 to 24, with higher scores indicating higher levels of dissociation.
Ketamine Side Effects - Mystical Experiences Questionnaire (MEQ) | 60 minutes after each treatment
  A 30-item questionnaire for participants to self-report the degree of dissociative and hallucinogenic experiences during the treatment. Each item is scored 0-5, with 0 indicating "none" and 5 indicating "extreme."
Ketamine Side Effects - Simulator Sickness Questionnaire | At baseline and 60 minutes after each treatment
  Tolerability of the VR experience will be assessed using the Simulator Sickness Questionnaire (SSQ). Participants will rate the degree to which they experienced 16 symptoms on a scale of 0 to 3, with 0 indicating "not at all" and 3 indicating "severe."
Cognitive Function - tele-MoCA | Baseline, 1 and 3 month follow-ups
  Any effect of ketamine and VR-K on cognitive function will be assessed using the telephone Montreal Cognitive Assessment (tele-MoCA). Scores range from 0 to 22, with higher scores indicating less cognitive impairment.
Change in EEG Metrics | Before, continuously during the 45-minute infusion, and up to 60 minutes after each treatment
  The effect of ketamine and VR-K on neural activity will be assessed using a Muse headband with advanced EEG brain sensors (https://ca.choosemuse.com/products/muse-2). Data will be collected using four EEG channels, two each on the anterior frontal (AF) and temporal-parietal (TP) regions, AF7, AF8, TP9, and TP10. Recordings will include data for five brainwaves: alpha, beta, delta, gamma, and theta. The change in EEG metrics will be assessed throughout each treatment and compared between the two treatment groups. Data will be collected using the Muse Lab software.
Patient Satisfaction - System Usability Scale | 60 minutes after the first and final VR-K treatments
  Participants in the VR-K group only will be asked to complete a VR system usability scale (VR-SUS) survey for VR technology to evaluate the ease of use of VR technology in this patient population. Participants will indicate their agreement with 8 statements on system usability on a scale of 1-5, with 1 indicating "strongly agree" and 5 indicating "strongly disagree."
Patient Satisfaction - Satisfaction Questionnaire | 60 minutes after the first and final VR-K treatments
  A satisfaction questionnaire surveying participants' subjective thoughts on the procedure experience. The questionnaire will ask participants' level of agreement with 12 statements regarding their experience (5-level scale, from "strongly agree" to "strongly disagree"), as well as ask about participants' preferences regarding video themes/features (open-ended questions).

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data will be made available upon reasonable request to study PI following publication of full trial results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This is a pilot trial and full inferential analysis will not be conducted until completion of the full trial. As such, data will be available following publication of the primary results of the subsequent full trial.
Access Criteria: Data and supporting information will be made available following reasonable request directly to study PI.